CLINICAL TRIAL: NCT02229643
Title: Neuroglobin and Nogo-A as Biomarkers for the Prognosis of Closed Traumatic Brain Injury
Brief Title: Serum Neuroglobin and Nogo-A Concentrations in Acute Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Chen, Doctor, Shanghai 6th People's Hospital
Other Study IDs: 658346
Record Dates: First submitted 2014-08-21; First posted 2014-09-01 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury; Neuroglobin; Nogo-A; Prognosis
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Traumatic brain injury: Patients delivered within 4 h whose highest abbreviated injury score (AIS) was 3 or less (other than head injury) were considered to be isolated traumatic brain injury cases and were included in this study.

SUMMARY:
Neuroglobin has been described as a marker of traumatic brain injury. Nogo-A plays an important role in mediating neuroanatomical plasticity and functional recovery following traumatic brain injury. The investigators sought to examine the changes in serum neuroglobin and Nogo-A concentrations in patients with traumatic brain injury during the initial 96-h posttraumatic period and assessed the relation of neuroglobin and Nogo-A to Glasgow Coma Score and prognosis of such patients with traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients who suffered head trauma and whose highest abbreviated injury score (AIS) was 3 or less (other than head injury)
* Patients who delivered to hospital within 4 h

Exclusion Criteria:

* Patients who suffered open injuries
* Patients who had existing prior neurological disease
* Patients whose serial serum samples could not be obtained
* Patients less than 18 years of age
* Patients who suffered severe life-threatening injury to organs other than the brain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient group comprised 21 male and 13 female. Their age ranged from 19 to 68 years, with mean age of 45.1 years. The mechanisms of trauma included motor vehicle collisions, falls, heavy strikes (patients who were hit by heavy objects such as bricks, sticks, or falling objects) and assaults. Types of lesions, as evidenced by radiologic and neurologic symptoms or signs, included cerebral contusions/lacerations, intracranial hematomas, brain stem injury and diffuse axonal injury.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Glasgow Outcome Scale scores | 6 months
  Glasgow Outcome Scale 1 = death; Glasgow Outcome Scale 2 = vegetative state; Glasgow Outcome Scale 3 = severe neurological deficit; Glasgow Outcome Scale 4 = mild neurological deficit and Glasgow Outcome Scale 5 = premorbid level of functioning or completely recovery. Unfavorable outcome was defined as a Glasgow Outcome Scale score of ≤ 3, and favorable outcome was defined as a Glasgow Outcome Scale score of > 3.

CONTACTS AND LOCATIONS:
Overall Officials: Lixia Xue, M.D., Ph.D., Study Director — Shanghai 6th People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China